CLINICAL TRIAL: NCT02032264
Title: Evaluation of the Efficacy of Next Generation Sequencing in Predicting Embryonic Karyotype and Subsequent Pregnancy Outcomes in in Vitro Fertilization Cycles (IVF)
Brief Title: Next Generation Sequencing Screening for Embryonic Ploidy Status
Acronym: nexgen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMA-2013-04
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: Next generation sequencing; Embryonic aneuploidy
MeSH Terms: conditions — Infertility | interventions — Prostaglandins D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive Chromosome Screening (Experimental): Trophectoderm biopsy will be performed on all blastocysts and CCS via next generation sequencing screening performed on biopsy samples. Patients will proceed with a single or double embryo transfer of the one or two morphologically best euploid embryos
  Interventions: Other: Comprehensive Chromosome Screening
- No Comprehensive Chromosome Screening (Placebo Comparator): The patients in this group will proceed with a single or double embryo transfer of the one or two morphologically best embryos.
  Interventions: Other: Morphologically Best

INTERVENTIONS:
Other: Comprehensive Chromosome Screening — On day 6 of embryo development, all embryos will undergo a trophectoderm biopsy using the standardized technique, as according to standard laboratory protocol and without regard to study. Comprehensive Chromosome Screening (CCS), will be performed via next generation sequencing and results will be available at the time of study completion.
  Other Names: PGD; CCS
  Arms: Comprehensive Chromosome Screening
Other: Morphologically Best — Patients in this arm of the study will not receive CCS in selection of their embryo for transfer. The best looking embryo (morphology) will be transferred
  Other Names: Unscreened; No CCS
  Arms: No Comprehensive Chromosome Screening

SUMMARY:
To evaluate the benefits of using next generation sequencing to assess embryonic aneuploidy. All viable blastocysts will be biopsied and cryopreserved for future transfer. After the final embryo is cryopreserved, patients will be randomized to either the intervention group or the control group. Patients and doctors are blinded to the randomization until study completion. A Double Embryo Transfer (DET) will be performed with either screened or unscreened embryos depending on randomization. A Single Embryo Transfer (SET) may occur in cases where only one embryo is available for transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IVF/CCS (no PGD banking)
* Patient meets ASRM guidelines for Double Embryo Transfer (DET)
* Donor Sperm OK
* AMH ≥ 1.2
* FSH ≤ 12
* BAFC ≥12
* Max 1 prior failed IVF cycle for patients 35-45 years old
* Patient <35 years old MUST have 1 prior failed IVF cycle

Exclusion Criteria:

* Chronic endometrial insufficiency
* Use of oocyte donor or gestational carriers
* Medical contraindications to Double Embryo Transfer (DET)
* Male Factor (<100,000 sperm or surgical sperm)
* Communicating hydrosalpinx (on HSG)
* Single gene disorders or sex selection

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Impact of next generation sequencing on the embryos produced from IVF on implantation rates | 2 years
  To evaluate the benefits, if any, of using next generation sequencing based Comprehensive Chromosome Screening (CCS) in the selection of embryos for transfer during clinical IVF cycles

SECONDARY OUTCOMES:
Delivery Rates | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, M.D., HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291
- [Derived] Tiegs AW, Tao X, Zhan Y, Whitehead C, Kim J, Hanson B, Osman E, Kim TJ, Patounakis G, Gutmann J, Castelbaum A, Seli E, Jalas C, Scott RT Jr. A multicenter, prospective, blinded, nonselection study evaluating the predictive value of an aneuploid diagnosis using a targeted next-generation sequencing-based preimplantation genetic testing for aneuploidy assay and impact of biopsy. Fertil Steril. 2021 Mar;115(3):627-637. doi: 10.1016/j.fertnstert.2020.07.052. Epub 2020 Aug 28. PMID 32863013